CLINICAL TRIAL: NCT01396408
Title: A Phase II Study of Sunitinib or Temsirolimus in Patients With Advanced Rare Tumours
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I206
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Advanced Rare Tumours
MeSH Terms: interventions — Sunitinib; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sunitinib (Active Comparator)
  Interventions: Drug: Sunitinib
- Temsirolimus (Active Comparator)
  Interventions: Drug: Temsirolimus

INTERVENTIONS:
Drug: Sunitinib — 50 mg PO daily for 28 days, q 6 weeks (1 cycle=6 weeks or 42 days)
  Arms: Sunitinib
Drug: Temsirolimus — 25 mg IV weekly (Days 1, 8, 15, 22, 29, 36), q 6 weeks (1 cycle=6 weeks or 42 days)
  Arms: Temsirolimus

SUMMARY:
This research is being done because there is no treatment that will cure this type of cancer. Although some types of chemotherapy can cause this cancer to shrink for a time, better options are needed.

DETAILED DESCRIPTION:
The purpose of this study is to find out what effects the study drugs - sunitinib or temsirolimus - will have on this type of cancer. The study will begin by finding out if sunitinib can shrink the cancer. If sunitinib does not work, temsirolimus will be tested next.

ELIGIBILITY:
Eligibility Criteria - ALL Patients

Patients must have histologically or cytologically confirmed diagnosis of a rare tumour as follows:

1. Vascular sarcomas: Angiosarcoma, hemangiosarcoma, hemangiopericytoma, hemangioblastomas;
2. Clear cell carcinomas of the ovary, endometrium;
3. Medullary thyroid carcinoma;
4. Neuroendocrine tumours: paragangliomas and pheochromocytomas only;
5. Adrenocorticocarcinoma;
6. Thymic carcinoma;
7. Fibrolamellar hepatocellular carcinoma;
8. Exploratory genetic cohort for sunitinib: Rare tumours with somatic or germline mutations in sunitinib targets such as VEGFR, PDGFR, KIT, RET;
9. Exploratory genetic cohort for temsirolimus: Rare tumours arising from known or suspected germline mutations in mTOR pathway such as PTEN, TS1/2, LKB1, NF1/2 or somatic mutations in the mTOR pathway such as mutation or amplification of P13K or AKT;
10. Unspecified cohort for exploratory evaluation. The unspecified histologies must also be rare tumours for which there are no traditional phase II clinical trials and for which there are clinical activity or laboratory data to support the likely sensitivity to the agents.
11. Ewing's Sarcoma Family of Tumours (ESFT) - relapsed or refractory.

    * Patients must have unresectable, locally advanced or metastatic disease for which there are no known life prolonging standard therapies.
    * Patients must have tumour tissue from their primary tumour available
    * Presence of clinically and/or radiologically documented disease. At least one site of disease must be unidimensionally measurable as follows:

    Chest x-ray ≥ 20 mm Ct scan (with slice thickness of ≤ 5 mm) - ≥ 10 mm --> Longest diameter Physical exam (using calipers) - ≥ 10 mm Lymph nodes by ct scan - ≥ 15 mm --> Measured in short axis

    All radiology studies must be performed within 21 days prior to registration (within 28 days if negative).
    * Age ≥ 16 years for cohorts #1-10; age ≥ 5 years for cohort #11 (ESFT) only.
    * Patients must have a life expectancy of at least 12 weeks.
    * ECOG performance status 0, 1 or 2.
    * Previous Therapy Chemotherapy: Patients may have received prior chemotherapy (no limit on number of prior regimens), however no prior treatment with relevant mTOR or VEGFR, KIT, RET, PDGFR inhibitors is permitted (i.e. to be eligible for sunitinib: no prior treatment with VEGFR, KIT, RET or PDGFR inhibitors permitted; to be eligible for temsirolimus: no prior treatment with mTOR inhibitors permitted). A minimum of 28 days (4 weeks) must have elapsed since the last dose of chemotherapy prior to registration. Patients must have recovered from any treatment related toxicities prior to registration.

    Radiation: Patients may have had prior radiation therapy. A minimum of 28 days (4 weeks) since the last dose of radiation must have elapsed prior to registration (exceptions may be made for low dose, palliative radiotherapy. Patients must have recovered from any acute toxic effects from radiation prior to registration.

    Previous surgery: is permitted provided that wound healing has occurred and at least 28 days have elapsed prior to registration if surgery was major.

    Laboratory Requirements:

    (must be done within 7 days prior to registration) Hematology Absolute granulocytes: ≥ 1.5 x 10^9/L Platelets: ≥ 100 x 10^9/L

    Chemistry:

    ALL Patients Bilirubin ≤ 1.5 x UNL (upper normal limit) AST and ALT ≤ 2.5 x UNL Serum Creatinine ≤UNL or: Creatinine clearance ≥ 60ml/min

    Chemistry:

    TEMSIROLIMUS Arm Only Fasting cholesterol ≤ 9.0 mmol/L Fasting triglycerides ≤ 4.56 mmol/L

    * Creatinine clearance to be measured directly by 24 hour urine sampling or as calculated by Cockcroft Formula: Females: GFR = 1.04 x (140-age) x weight in kg serum creatinine in μmol/L Males: GFR = 1.23 x (140-age) x weight in kg serum creatinine in μmol/L
    * Patient or guardian consent must be obtained on all patients according to local Institutional and/or University Human Experimentation Committee requirements. Children > 8 years old whose parent or guardian has signed consent on their behalf may also sign assent if desired. It will be the responsibility of the local participating investigators to obtain the necessary local clearance, and to indicate in writing to the NCIC CTG Study Coordinator that such clearance has been obtained, before the trial can commence in that centre. Because of differing requirements, a standard consent form for the trial will not be provided but a sample form is provided. A copy of the initial full board REB approval and approved consent form must be sent to the central office. The patient or their parent/legal guardian must sign the consent form prior to registration. Please note that the consent form for this study must contain a statement which gives permission for the NCIC CTG and monitoring agencies to review patient records.
    * Patients must be accessible for treatment, response assessment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial. (Call the NCIC CTG office at 613-533-6430 if questions arise regarding the interpretation of this criterion.) Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.

    In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient registration.

    Ineligibility Criteria - ALL Patients

    Patients who fulfill any of the following criteria are not eligible for admission to either the sunitinib treatment arm (Arm A) or temsirolimus arm (Arm B) of this study:
    * Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer or other solid tumours curatively treated with no evidence of disease for ≥ 3 years.
    * Patients who have had prior treatment with relevant mTOR or VEGFR, KIT, RET, PDGFR inhibitors. Patients who have had prior treatment with mTOR inhibitors are ineligible for temsirolimus; patients who have had prior treatment with VEGFR, KIT, RET or PDGFR inhibitors are ineligible for sunitinib.
    * Pregnant or lactating women. Women of childbearing potential must have a urine pregnancy test proven negative within 7 days prior to registration. Men and women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
    * Patients with known symptomatic brain metastases (a brain CT is not necessary to rule out brain metastases, unless there is clinical suspicion of CNS involvement). Patients with treated and radiologic or clinical evidence of stable brain metastases, with no evidence of cavitation or hemorrhage in the brain lesion, are eligible providing that they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 1 week prior to entry).
    * Patients with known hypersensitivity to the relevant study drug or its components, or compounds of similar chemical or biologic composition.
    * Patients receiving concurrent treatment with other anti-cancer therapy or other investigational agents.
    * Patients with serious illness or medical condition which would not permit the patient to be managed according to the protocol including, but not limited to:

      1. History of significant neurologic or psychiatric disorder which would impair the ability to obtain consent or limit compliance with study requirements
      2. Active uncontrolled infection
      3. Any other medical conditions that might be aggravated by treatment
      4. Serious or non-healing wound, ulcer, or bone fracture.
      5. Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment. Patients believed to be at high risk for fistula formation because of the location and extent of their disease should not be enrolled.

    Ineligibility Criteria - SUNITINIB Arm Only

    Patients who fulfill any of the following criteria are not eligible for admission to the sunitinib treatment arm (Arm A) of this study:
    * Patients with pre-existing cardiovascular conditions and/or symptomatic cardiac dysfunction as follows:

      1. QTc prolongation (defined as a QTc interval equal to or greater than 500 msec) or other significant abnormalities on screening ECG (required within 14 days prior to registration).
      2. Current or history of Class III or IV heart failure as defined by the NYHA functional classification system.
      3. Patients with prior anthracycline exposure, previous central thoracic radiation that included heart in radiation port, or a history of NYHA Class II cardiac function UNLESS they are currently asymptomatic with respect to cardiac function AND left ventricular ejection fraction (LVEF) > lower limit of normal (LLN) of institution as assessed by screening MUGA or ECHO (required within 14 days prior to registration).
      4. Poorly controlled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg.
      5. Myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry
      6. History of pulmonary embolism within the past 12 months; patients with incidental pulmonary emboli found on routine scanning > 6 months prior to registration may be eligible.
      7. History of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry.
    * Patients who require use of therapeutic doses of coumadin-derivative anticoagulants such as warfarin are excluded, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis. Use of low molecular weight heparin is permitted provided the patient's INR is ≤ 1.5. INR on screening coagulation (required within 7 days prior to registration).
    * Patients with bowel obstruction or GI tract disease resulting in an inability to absorb oral medication , such as uncontrolled inflammatory GI disease (e.g. Crohn's disease, ulcerative colitis) or post surgical malabsorption characterized by uncontrolled diarrhea that results in weight loss and vitamin deficiency or requires IV hyperalimentation; or any condition that would preclude compliance with oral medication.
    * Patients with pre-existing hypothyroidism are ineligible, unless they are euthyroid on medication.
    * Inability to discontinue drugs known to be potent inhibitors or inducers of cytochrome P450 (CYP3A4). Patients must be off these medications 7-12 days prior to the first dose of sunitinib.

    Inhibitors- prohibited 7 days before dosing and during study. azole antifungals (ketoconazole, itraconazole, miconazole, fluconazole) HIV protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfinavir) clarithromycin verapamil erythromycin delavirdine diltiazem nefazodone telithromycin

    Inducers- prohibited 12 days before dosing and during study. rifampin phenytoin rifabutin St. John's wort carbamazepine efavirenz phenobarbital tipranavir

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2012-02-09 (Actual); Primary Completion 2015-07-06 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response | Every 4 weeks
  Objective response as assessed by RECIST version 1.1 criteria as a 30% decrease in the sum of the longest diameters of the target lesions (partial response) maintained for at least 4 weeks, or complete disappearance of disease and cancer related symptoms (complete response), also maintained for at least 4 weeks. Early progression is defined as progressive disease at or prior to the first assessment. The 95% confidence interval for response rate will be calculated. The median and range of the duration of response will be assessed

SECONDARY OUTCOMES:
Efficacy Outcomes | 48 months
  * Response duration: median and range
  * Time to progression: median, 95% confidence interval
  * Progression free survival: median, 95% confidence interval
  * Overall survival: median, 95% confidence interval
  * Comparison of the time to first and second progression for patients who receive sunitinib and temsirolimus in sequence.
Translational Research | 48 months
  Primary tumour tissue specimens and baseline blood samples, will be obtained from all subjects prior to first dose for genetic analysis and other evaluation. In addition, optional for responding patients will be a fresh tumour biopsy at time of progression and also optional for patients entered in the second stage of accrual for any disease cohort will be fresh tumour biopsy at baseline.
Safety Monitoring | Daily up to an expected average of 4 weeks after treatment
  Adverse events will be monitored on an ongoing basis by the central office and their frequencies reported annually at investigators' meetings.

CONTACTS AND LOCATIONS:
Overall Officials: Hal Hirte, Study Chair — Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, ON Canada
Locations (17):
- Canada (17):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Izaak Walton Killam (IWK) Health Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No